CLINICAL TRIAL: NCT00466232
Title: Phase I Study of Weekly Topotecan in Combination With Sorafenib in Treatment of Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3557-07-C
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2007-04

CONDITIONS: Small Cell Carcinoma; Lung Cancer
Keywords: Small Cell; Lung Cancer; Treatment
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms | interventions — Topotecan; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Weekly Topetecan in combination with Sorafenib
  Interventions: Drug: Topotecan; Drug: Sorafenib

INTERVENTIONS:
Drug: Topotecan — 4 mg/m2 IV on day 1, 8, 15. Repeat every 28 days.
  Other Names: Hycamtin
Drug: Sorafenib — Dose escalation study at 3 dose levels: 200 mg po daily, 200 mg po bid, 400 mg po bid.
  Other Names: Nexavar

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose of sorafenib up to the full active dose when combined with standard weekly dosing of topotecan in patients with recurrent small cell lung cancer and to characterize the toxicities associated with the combination of topotecan and sorafenib in this patient population

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) comprises approximately 15 percent of all lung cancers in the United States. It is highly correlated with tobacco use and occurs almost exclusively in smokers. SCLC is a particularly virulent malignancy characterized by rapid growth and a tendency to metastasize early in the disease course. In first line treatment, SCLC has a high response rate to cytotoxic chemotherapy. Unfortunately, the disease develops drug resistance in almost all cases resulting in recurrence. In second line treatment, the likelihood of response to treatment is considerably less. Multiple agents have been used in this setting with response rates typically around 25% and median survival of less than 6 months1-3. There is clearly a great need for more effective treatments in this disease.

Topotecan is a semi-synthetic, water soluble derivative of camptothecin, a cytotoxic alkaloid extracted from plants of the genus Camptotheca. Its mechanism of action is inhibition of topoisomerase I, an enzyme necessary to relieve torsional strain of DNA which is necessary to carry out replication. This results in DNA double-strand breaks and ultimately cell death. Topotecan has demonstrated activity in a number of malignancies and is currently indicated for the treatment of ovarian cancer, cervical cancer and recurrent small cell lung cancer.

Topotecan has demonstrated single agent activity in recurrent small cell lung cancer in a number of trials. Reported response rates range from 2 to 31%3-7. A phase III trial compared topotecan to CAV (cyclophosphamide, doxorubicin and vincristine) in treatment of recurrent SCLC5. Response rate, survival and time to progression were similar in both groups. The topotecan group demonstrated significant improvement in symptoms including anorexia, fatigue and dyspnea. This led to FDA approval of topotecan for treatment of recurrent SCLC.

The dose limiting toxicity of topotecan is hematologic. The approved schedule of administration is 1.5mg/m2 daily x 5 every 21 days. A modified schedule of weekly administration at 4mg/m2 has been shown to have similar efficacy with less toxicity8 and has been widely adopted in clinical practice.

Sorafenib is an oral multi-kinase inhibitor with effects on tumor proliferation and tumor angiogenesis. It has several biochemically important mechanisms including inhibition of Raf-1 and B-Raf which are pivotal components of the Ras/Raf/Mek/Erk signaling pathway. It also has inhibitory activity against the tyrosine kinases for VEGF and PDGFR as well as Flt-3 and c-kit.

Sorafenib has been safely combined with full dose cytotoxic chemotherapy in several Phase I trials9-11. There is no data on the combination of topotecan and sorafenib to date. Sorafenib is metabolized in the liver undergoing oxidation via CYP3A4 and glucuronidation via UGT1A9. There is no evidence that topotecan affects activity of the cytochrome P450 pathways suggesting low likelihood of a drug-drug interaction. There are no significant overlapping toxicities making this an ideal drug combination to investigate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven small cell carcinoma of bronchogenic origin.
* Must have received one course of systemic chemotherapy which included cisplatin or carboplatin. Chemotherapy administered during radiation is allowable.
* Must have radiographically documented disease recurrence or progression by CT scan or bone scan. CNS only recurrence is not sufficient. Measurable disease per RECIST criteria is not required.
* ECOG Performance status of 0 to 2
* Adequate organ function within 14 days of study enrollment as defined by the following:

  * Absolute neutrophil count ≥ 1500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 gm/dL
  * Creatinine ≤ 1.5 mg/dL
  * Bilirubin < 1.5 times upper limit of normal (x UNL)
  * Alkaline phosphatase, aspartate transaminase and alanine transaminase < 3 x ULN (may be <5 x ULN if hepatic metastases)
* Women of childbearing potential and sexually active males must use an effective method of contraception during the study and for 3 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Treated brain metastases that are stable for a minimum of 4 weeks following surgery or radiation and off therapeutic glucocorticoids are allowed.
* INR<1.5 or a PT/PTT within normal limits. Patients receiving anti- coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Pregnant or breast feeding.
* Myocardial infarction or cerebrovascular accident within 6 months.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg despite optimal medical management.
* History of other active invasive malignancy (except for basal cell or squamous cell skin cancer) within 12 months.
* Major surgery within 4 weeks.
* Chemotherapy within 4 weeks.
* Cardiac disease: Congestive heart failure > NYHA Class II, unstable or new-onset angina within prior 3 months.
* History of bleeding diathesis or coagulopathy.
* Active clinically serious infection > CTCAE Grade 2.
* Ventricular arrhythmias requiring anti-arrhythmic therapy.
* Serious non-healing wound, ulcer or fracture.
* Any hemorrhage or bleeding event > CTCAE Grade 3 within 4 weeks of study enrollment.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Known human immunodeficiency virus (HIV) or chronic hepatitis B or C infection.
* Any condition that impairs patient's ability to swallow whole pills.
* Any gastrointestinal malabsorption syndrome
* Use of St. John's wort or rifampin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the maximum tolerated dose of sorafenib up to the full active dose when combined with standard weekly dosing of topotecan in patients with recurrent small cell lung cancer and to | 2 years
characterize the toxicities associated with the combination of topotecan and sorafenib in this patient population | 2 years

SECONDARY OUTCOMES:
To evaluate the objective response rate (CR, PR or stable disease) | 2 years
To measure time-to-event efficacy looking at the following variables: | 2 years
o Time to disease progression | 2 years
o Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leach, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Park Nicollet Institute, Saint Louis Park, Minnesota, United States